CLINICAL TRIAL: NCT04269967
Title: A Pilot Feasibility Study of a Tele-rehabilitation System Among Women Who Undergo a Unilateral Mastectomy for Breast Cancer
Brief Title: A Pilot Tele-rehabilitation Trial for Breast Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Singapore General Hospital (Other); National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Miho Asano, Assistant Professor, National University of Singapore
Other Study IDs: 2019/00283
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tele-rehabilitation: Patients who choose tele-rehabilitation
  Interventions: Other: Receiving routine rehabilitation care via tele-rehabilitation system
- Usual care: Patients who choose usual (rehabilitation) care

INTERVENTIONS:
Other: Receiving routine rehabilitation care via tele-rehabilitation system — Drain care education, self-massage techniques and exercise (PT and OT)
  Groups: Tele-rehabilitation

SUMMARY:
Breast cancer is the leading cancer affecting women in Singapore. Breast cancer survivors commonly experience declined physical function and quality of life, due to their upper limb morbidity and wound issues post-surgery. Rehabilitation therapy can address the aforementioned issues that the survivors may experience during their recovery. No therapy however, can be effective if patients do not utilize them. Home-based telehealth (e.g., tele-rehabilitation) self-managed by patients and guided by healthcare professionals can potentially improve the service use and recovery. This study aims to understand the lived experience of post-mastectomy tele-rehabilitation and recovery process among female patients who undergo a unilateral mastectomy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female 21 years and over
* Underwent a recent unilateral breast surgery (wide excision or simple mastectomy) with lymph nodes removed
* Speak and write English or Mandarin;
* No psychiatric history or chronic psychiatric condition as assessed by referring clinician

Exclusion Criteria:

* Having breast reconstruction
* Having legal blindness or severe visual impairment
* Having life expectancy of less than three months (12- weeks)
* Having previous upper limb injury or conditions that limit passive ranges of shoulder flexion (<150°), elbow extension/flexion (0/145°)

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females identified by their healthcare providers.
Study Population: Adults female who are undergoing or underwent a unilateral breast surgery (wide excision or simple mastectomy) with lymph nodes removed at two participating sites in Singapore.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The experience of rehabilitation (i.e., drain care, exercise and massage) | 12 weeks from the baseline assessment
  We will interview our participants about their experience of going through a rehabilitation process. This is qualitative data.
Shoulder range of motion | Pre rehabilitation (week 0) and post-rehabilitation (week 12)
  Shoulder ranger of motion will be measured in degree.
Arm circumference | Pre rehabilitation (week 0) and post-rehabilitation (week 12)
  Arm circumference will be measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: Miho Asano, Principal Investigator — SSHSPH NUS
Locations (1):
- Miho Asano, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asano M, Koh GC, Madhukumar P, Teng GYH, Liew PLL, Nagalingam S, Tan MLM, Ng YS, Tan BKT. Study protocol: a pilot quasi-experimental trial of tele-rehabilitation and tele-drain care post-mastectomy. Pilot Feasibility Stud. 2021 Feb 1;7(1):39. doi: 10.1186/s40814-021-00776-5. PMID 33522962